CLINICAL TRIAL: NCT06452420
Title: The Degree of Knowledge and Attitude of Medical Residents and Interns in Egypt Regarding Emergency Treatment of Traumatic Dental Injuries
Brief Title: Knowledge and Attitude of Medical Residents and Interns in Egypt Regarding Traumatic Dental Injuries
Status: Not yet recruiting | Type: Observational
Sponsor: Ghada Sayed Ahmed Sayeh (Other)
Responsible Party: Sponsor-Investigator, Ghada Sayed Ahmed Sayeh, Principal investigator, Cairo University
Organization: Cairo University (Other)
Other Study IDs: QuestionnareTDI
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Traumatic Dental Occlusion
Keywords: Traumatic Dental Injuries
MeSH Terms: conditions — Dental Occlusion, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Traumatic dental injuries — The Degree of knowledge and Attitude of Medical Residents and Interns in Egypt regarding Emergency treatment of traumatic dental injuries.

SUMMARY:
Aim of the study This study intends to evaluate medical residents and interns fundamental knowledge and attitude regarding the management of TDIs in Egypt.

DETAILED DESCRIPTION:
II. Introduction:

Scientific background:

Statement of the problem Violence, sports, auto accidents and falls are the most frequent causes of traumatic dental injuries (TDIs), which are regarded as the most serious oral health issue affecting children. It has been reported that physicians are the first who assist patients with TDIs. In hospitals, patients typically anticipate receiving care from emergency department doctors. Thus, before referring patients to a dentist for follow-up care, physicians are typically obliged to handle the emergency therapy phase and stabilize acute TDIs.

Global studies found that pediatricians and even emergency room doctors lacked the knowledge to manage TDIs. This might be explained that emergency room doctors might not believe that dental emergencies are one of the responsibilities of the emergency room staff. Thus proposed changing the medical curricula to include more knowledge and expertise for the management of TDIs.

The knowledge and attitude of medical residents and interns who will treat TDIs should be evaluated. However, multiple studies have found that medical students had little awareness of TDIs, with the majority of them (between 70 and 90 percent) claiming that their undergraduate curricula did not include any formal instruction in TDIs. Additionally, the majority of students felt that understanding TDIs was not essential for their future employment.

Review of literature:

Dental traumatology includes the study of acute dental trauma involving injury to the teeth, gums, and jaw bones. Children and adolescents frequently sustain dental injuries, which is considered to be a serious public dental health issue. Traumatic dental injuries are considered the second most common dental issue worldwide, with dental caries being the first, with a frequency of permanent dentition of 15.2% and primary dentition of 22.7%.

According to reports, dental trauma occurs more frequently than non-oral traumas, especially in the first 10 years of life. In Egypt, the prevalence of traumatic dental injuries represents 10% for primary dentition and 14.6% in permanent dentition. Traumatic dental injury (TDI) is an impact injury to the teeth and/or supporting tissues that can be accidental or purposeful. It cannot be anticipated and frequently requires emergency care due to its nature. Although it can happen at any age, the majority of TDI occurs in children.

According to literature reviews, between one-third and one-fourth of kids in the primary dentition age range experience TDIs. Parents and kids may find this issue upsetting, and it may also have negative psychological, aesthetic, and bodily effects Dental trauma is frequently linked to sports, falls, and collisions with persons or objects, all of which are frequent occurrences in children's daily lives. The primary location for TDI is at home, followed by preschool or school and outside.

The two steps of the treatment for TDIs are immediate emergency care and follow-up. To reduce the possibility of short-term and long-term negative outcomes, proper care must be provided during the whole treatment process. Dental trauma therapy is crucial in the short term to contract the pain, restore oral function and appearance, decrease dental anxiety and prevent infections.

A lack of knowledge regarding such injuries and the con- sequent failure to provide adequate treatment may lead to functional deficits and aesthetic defects, especially in growing patients. As a result, articles published in the literature of the last five years on the prevention, first aid and certification of dental trauma in children have been considered. It's crucial for medical professionals working in hospital emergency rooms to be knowledgeable about and efficient in treating TDI. It is essential for medical professionals to be able to provide adequate and appropriate emergency care to stabilize dental injuries and dramatically increase the survival rate of the affected tooth because the majority of TDI victims present to emergency departments or general medical practice surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Positive subject acceptance for participation in the study
* Medical interns and residents who work in Surgery, Paediatrics and Emergency departments.
* Both genders.

Exclusion Criteria:

* Medical residents and interns who refuse to participate.
* Medical interns and residents who don't use social networks

Ages: 24 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: Age: 24-30 Years Gender: Male /female Educational level: Medical residents and interns
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The degree of knowledge and attitude of medical residents and interns in Egypt regarding emergency treatment of traumatic dental injuries. | Baseline
  outcome: Degree of knowledge and attitude of medical residents and interns in Egypt regarding emergency treatment of traumatic dental injuries.
  Measurement method:
  Questionnaire
  Unite of measurement:
  Binary question (yes/no) Multiple choice question.

CONTACTS AND LOCATIONS:
Overall Officials: shereen bader, Doctor, Principal Investigator — Cairo U

REFERENCES:
- [Background] Ishida Y, Watanabe K, Kobayashi S, Kihar M. Selective alpha-adrenoceptor blocking actions of a new derivative of 2-halogenotheylamine: 6-(2-bromoethyl)-10,11-methylenedioxy-5,6,7,8-tetrahydrodibenz[c,e]azocine. Jpn J Pharmacol. 1976 Oct;26(5):607-14. doi: 10.1254/jjp.26.607. PMID 12395